CLINICAL TRIAL: NCT04633941
Title: Comparing the Impact of Social Distancing and Lockdown on Bariatric Patients Versus Non-Surgical Obese Patients During COVID-19 Pandemic - Cross Sectional Study
Brief Title: Impact of Social Distancing on Bariatric Versus Non-Surgical Obese Patients During COVID-19 Pandemic
Status: Completed | Type: Observational
Sponsor: Singapore General Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: HenryLew
Record Dates: First submitted 2020-11-12; First posted 2020-11-18 (Actual); Last update posted 2020-11-20 (Actual); Status verified 2020-11

CONDITIONS: Diabetes Mellitus, Type 2; Obesity, Morbid; Bariatric Surgery Candidate
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Obesity, Morbid | interventions — Standard of Care

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Post Bariatric Surgery: Post Bariatric Surgery more than 6 month. Obesity (BMI 30 kg/m2 and above), English literate and having mental capacity to make their own decisions. Patients were excluded if they had undergone bariatric surgery ≤ 6 months ago, have active eating disorders, are pregnant or had given birth ≤ 6 months ago. Patients who were admitted to hospital or tested positive for COVID-19 were excluded too. Patients who had symptoms of active severe psychological and psychiatric conditions like psychosis, self-harm, suicide, hallucinations were also excluded
  Interventions: Other: Standard Care
- Medical Weight Management: Obesity (BMI 30 kg/m2 and above), English literate and having mental capacity to make their own decisions. Patients were excluded if they had undergone bariatric surgery ≤ 6 months ago, have active eating disorders, are pregnant or had given birth ≤ 6 months ago. Patients who were admitted to hospital or tested positive for COVID-19 were excluded too. Patients who had symptoms of active severe psychological and psychiatric conditions like psychosis, self-harm, suicide, hallucinations were also excluded
  Interventions: Other: Standard Care

INTERVENTIONS:
Other: Standard Care — Standard Care

SUMMARY:
In response to the COVID-19 pandemic, weight management programs and metabolic surgery have been deferred to contain the virus. Quarantine and social distancing negatively impact dietary, exercise and psychological health of obese individuals. The study aims to evaluate the impact of social distancing measures on post-metabolic surgery patients compare to non-surgical obese patients and discuss potential strategies for management post COVID-19.

DETAILED DESCRIPTION:
In Singapore, a nationwide partial lockdown, termed the "circuit breaker" was imposed from 7th April until 1st June 2020 in response to the COVID-19 pandemic (Appendix A). Our study aims to evaluate the impact of social distancing and lockdowns during this circuit breaker period on our patients with obesity, either post-metabolic surgery (MS) or undergoing active medical management (MM), during the COVID-19 pandemic in Singapore. Results will help inform and address the challenges in patient care that this pandemic has brought to light, its long-term implications on the management of the bariatric patient and discuss potential strategies for the management of a bariatric patient in a post COVID-19 society. To the knowledge of this paper, this is the first study to compare the impact of COVID on MS and MM patients which will allow understanding of unique stressors faced by MS patients

This study adopted a cross-sectional survey design to evaluate the impact of lockdown social distancing measures on obese patients in Singapore. The study conducted either face-to-face questionnaires in the clinic after lockdown for those who were not suitable for video consultation or questionnaires administered via telecommunication channels such as WhatsApp

ELIGIBILITY:
Inclusion Criteria:

* Obesity (BMI 30 kg/m2 and above)
* English literate
* Mental capacity to make their own decisions

Exclusion Criteria:

* Undergone bariatric surgery ≤ 6 months ago
* Have active eating disorders
* Pregnant or had given birth ≤ 6 months ago
* Admitted to hospital or tested positive for COVID-19
* Exhibit symptoms of active severe psychological and psychiatric conditions like psychosis, self-harm, suicide, hallucinations that may hinder them from providing accurate responses.

Ages: 18 Years to 65 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients with obesity, either post-metabolic surgery (MS) or undergoing active medical management (MM), during the COVID-19 pandemic in Singapore
Sampling Method: Non-Probability Sample
Enrollment: 272 (Actual)
Dates: Start 2020-06-01 (Actual); Primary Completion 2020-07-30 (Actual); Study Completion 2020-07-30 (Actual)

PRIMARY OUTCOMES:
Weight | June2020-July2020
  1 question asked about participants weight in kg before the lockdown; 1 question asked participants about weight in kg during lockdown

SECONDARY OUTCOMES:
Blood Sugar Control | June2020-July 2020
  Participants were asked 1 question on how well blood sugar was controlled before the lock down. An ordinal scale was used: Very Poor, Poor, Reasonable, Good, Very Good. Participants were asked 1 question on how well blood sugar was controlled during the lock down. An ordinal scale was used: Very Poor, Poor, Reasonable, Good, Very Good.
Medical Adherence | June 2020-July2020
  Participants were asked how often medication was missed before the lockdown with1 question using an ordinal scale: Never, Once in a while, Sometime, Usually, All the Time. Participants were asked how often medication was missed during the lockdown with1 question using an ordinal scale: Never, Once in a while, Sometime, Usually, All the Time.
Stress level | June 2020-July2020
  Participants were asked on the level of stress before the lockdown using a Likert scale of 1-10; with 1=not stressful at all; 10= extremely stressful. Participants were asked level of stress were during the lockdown using a Likert scale of 1-10; with 1=not stressful at all; 10= extremely stressful.
Physical Activity Level | June2020-July 2020
  Participants were asked frequency of exercise before the lockdown on a ordinal scale ranging from less than 1 time a week; Once a week; 2-3 times a week;4-5 times a week; More than 5 times a week. Participants were asked frequency of exercise during the lockdown on a ordinal scale ranging from less than 1 time a week; Once a week; 2-3 times a week;4-5 times a week; More than 5 times a week

CONTACTS AND LOCATIONS:
Overall Officials: Chin Hong Lim, FRCS, Principal Investigator — Staff
Locations (1):
- Singapore General Hospital, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: No